CLINICAL TRIAL: NCT02523027
Title: Oral Nutritional Supplementation in Picky Eating Children
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Abbott Nutrition (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: DA11
Record Dates: First submitted 2015-08-12; First posted 2015-08-14 (Estimated); Last update posted 2018-03-14 (Actual); Status verified 2018-03

CONDITIONS: Children - Malnutrition
MeSH Terms: conditions — Child Nutrition Disorders | interventions — Dietary Supplements

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental Group 1: (Experimental): Oral nutritional supplement (List No S691/Z0) and dietary counseling
  Interventions: Dietary Supplement: Oral nutritional supplement (List No S691/Z0); Other: Dietary Counselling
- Experimental Group 2 (Experimental): Oral nutritional supplement (List No- P968/Z0) and dietary counseling.
  Interventions: Dietary Supplement: Oral nutritional supplement; Other: Dietary Counselling
- Control Group (No Intervention): Dietary Counselling only.

INTERVENTIONS:
Dietary Supplement: Oral nutritional supplement (List No S691/Z0) — (List No S691/Z0)
  Arms: Experimental Group 1:
Dietary Supplement: Oral nutritional supplement — (List No- P968/Z0)
  Arms: Experimental Group 2
Other: Dietary Counselling — Regular dietary counseling conducted by a trained hospital dietitian.
  Arms: Experimental Group 1:; Experimental Group 2

SUMMARY:
This study will investigate the effect of two oral nutritional supplements (ONS) along with dietary counseling vs dietary counseling alone on growth among picky eating children from India, aged > 24 months to ≤ 48 months over a period of 90 days.

DETAILED DESCRIPTION:
Study Objective:

To investigate the effect of two oral nutritional supplements (ONS) along with dietary counseling vs dietary counseling alone on growth among picky eating children from India, aged > 24 months to ≤ 48 months over a period of 90 days.

Number of Subjects / Length of Participation:

Approximately 321 subjects (107 subjects per group) will be enrolled from estimated 8-10 study centers to obtain at least 255 evaluable subjects (85 subjects per group), assuming 20% attrition rate. Expected total duration for the study is approximately 12 months.

Study Design :

* Prospective, randomized, double blinded study, with two parallel treatment groups and an open-labeled control group multicenter clinical study Eligible subjects will be randomized into three groups
* Experimental Group 1: Oral nutritional supplement and dietary counseling. (List No S691/Z0)
* Experimental Group 2: Oral nutritional supplement and dietary counseling. (List No- P968/Z0)
* Control Group: Dietary counseling.

ELIGIBILITY:
Inclusion Criteria:

1. Child is > 24 months and ≤ 48 months of age at visit 1.
2. Child of either gender (Male and Female).
3. Child has a weight-for-height between 3rd - 15th percentiles according to current WHO Growth Charts at visit 1. (WHO Growth Chart 2007)
4. Child is a picky eater, defined as meeting at least two of the following criteria. A child, who:

   * eats only a limited number of foods
   * is unwilling to try new foods
   * refuses to eat vegetables and/or foods from other food groups
   * shows strong food likes and dislikes
   * has behaviors that disrupt mealtime
5. Child is a habitual milk drinker at least 1 glass (approximately 200mL) of milk daily.
6. Child is able to consume foods and beverages orally.
7. Child's Legal Guardian (LG) or parent(s) is willing to abstain from giving additional non-study nutritional supplements including vitamin/mineral supplements, micronutrient fortified beverages, oral nutritional supplements other than the study product during the study intervention period.
8. Child's Legal Guardian (LG) or parent(s) has voluntarily signed and dated an informed consent form (ICF), approved by an Independent Ethics Committee/Institutional Review Board (IEC/IRB) prior to any participation in the study.
9. Child's Legal Guardian (LG) or parent(s) is able and willing to follow study procedures and record data in parent diary and complete any forms or assessments needed throughout the study.
10. Child's Legal Guardian (LG) or parent(s)is not planning to relocate during the study period

Exclusion Criteria:

1. Child has been diagnosed with Lactose Intolerance & Galactosemia according to medical records or Legal Guardian (LG) /parent report.
2. Child has been diagnosed or is known to be allergic or intolerant to any ingredient found in the study product according to medical records or Legal Guardian (LG)/parent report.
3. Child has a current acute or chronic infection including respiratory infection, diarrhea, acute or chronic, Hepatitis B or C, HIV infection or tuberculosis according to medical records or Legal Guardian (LG)/parent report.
4. Child has been diagnosed with presence of severe gastrointestinal disorders including celiac disease, short bowel syndrome, pancreatic insufficiency, or cystic fibrosis according to medical records or Legal Guardian (LG)/parent report.
5. Child has been diagnosed with neoplastic, renal, hepatic or cardiovascular disease according to medical records or Legal Guardian (LG) /parent report.
6. Child has been diagnosed with hormonal or metabolic disorders according to medical records or Legal Guardian (LG) /parent report.
7. Child has been diagnosed with congenital disease or genetic disorders such as atrial or ventricular wall defects, or Down's syndrome according to medical records or Legal Guardian (LG) /parent report.
8. Child has been diagnosed with infantile anorexia nervosa according to medical records or Legal Guardian (LG) /parent report.
9. Child has been diagnosed with a developmental disability, including physical disorders such as cerebral palsy, or developmental delay according to medical records or Legal Guardian (LG) /parent report.
10. Child has been diagnosed with disorders of hemoglobin structure, function or synthesis according to medical records or Legal Guardian (LG) /parent report.
11. Child has a clinically significant nutritional deficiency requiring specific treatment with another nutritional supplement (other than the study product) as diagnosed by the investigator.
12. Child has any other clinically significant medical condition, which in the investigator's opinion, makes him or her unsuitable for inclusion in the study.

Ages: 2 Years to 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 321 (Actual)
Dates: Start 2016-06-21 (Actual); Primary Completion 2017-02-17 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Change in WHO weight-for-height percentile | Day 1 to Day 90

SECONDARY OUTCOMES:
Change in weight-for-height WHO z-score | Day 1 to Day 90
Change in weight-for-age WHO z-score and percentile | Day 1 to Day 90
Change in height-for-age WHO z-score and percentile | Day 1 to Day 90
Change in BMI-for-age WHO z-score and percentile | Day 1 to Day 90
Change in Mid Upper Arm Circumference-for-age WHO z-score and percentile | Day 1 to Day 90
Average energy macronutrients (Carbohydrates, Fats, & Proteins) and micronutrients consumption via 24 hr dietary recall | Days 1, 7, 30, 60 and 90
Change in appetite score | Days 1, 7, 30, 60 and 90
Palatability scores for the oral nutritional supplements | Days 7, 30, 60 and 90
Change in weight-for-height WHO z-score and percentile | Day 1 to Day 90
Average energy macronutrients (Carbohydrates, Fats, & Proteins) and micronutrients consumption via 24 hr dietary recall | Day 1, 7, 30, 60 and 90

CONTACTS AND LOCATIONS:
Overall Officials: Irfan Shaikh, M.D., Study Chair — Abbott Nutrition
Locations (11):
- India (11):
  - Praveen Cardiac Centre, Vijayawada, Andhra Pradesh
  - St. Theresa's Hospital, Hyderabad, Erragadda, Sanath Nagar
  - Sangini Hospital, Ahmedabad, Gujarat
  - JSS Medical College & Hospital, Mysore, Karnataka
  - Jehangir Clinical Development Centre, Jehangir Hospital, Pune, Maharashtra
  - Medipoint Hospitals, Pune, Maharashtra
  - Noble Hospital, Pune, Maharashtra
  - Sterling Multispeciality Hospital, Pune, Maharashtra
  - Kanchi Kamakoti Child Trust Hospital, Chennai, Tamil Nadu
  - Ajanta Research Centre, Ajanta Hospital & IVF Centre, Lucknow, Uttar Pradesh
  - Institute of Child Health, Kolkata, West Bengal

IPD SHARING:
Plan to Share IPD: No